CLINICAL TRIAL: NCT00893568
Title: Post Traumatic Stress Disorder and Neural Mechanisms Involved in Its Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2009/01; 2009-A00193-54
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Post Traumatic Stress Disorders
Keywords: Post traumatic stress disorder PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy volunteers (Active Comparator): Healthy volunteers without treatment
  Interventions: Other: resonance magnetic imaging (fMRI),
- CBT (Experimental): Psychotraumatized patients treated by Cognitive and Behavioral Therapies (CBT)
  Interventions: Other: resonance magnetic imaging (fMRI),
- EMDR (Experimental): Psychotraumatized patients treated by Eye Movement Desensitization and Reprocessing (EMDR)
  Interventions: Other: resonance magnetic imaging (fMRI),

INTERVENTIONS:
Other: resonance magnetic imaging (fMRI), — a cerebral study will be performed at the neuroanatomic and functional levels by resonance magnetic imaging (fMRI) realized in three times (before, one week and six months after treatment)

SUMMARY:
The post traumatic stress disorder PTSD arises when the physiological response to stress does not come to its term. This study aims to explore the cognitive, psycho physiological and cerebral mechanisms involved in PTSD, in fear conditioning and face matching tasks, before and after treatment.PTSD patients will be recruited by Pr Jean-Claude Samuelian in his service at the Conception Hospital and by Pr Jean-Michel Azorin in his service at the Sainte Marguerite Hospital (Marseille) and will undergo either CBT or EMDR within those same services. The tasks they will be asked to perform will study the psycho physiological, cognitive and central mechanisms involved in PTSD and its treatment. All in all, 17 healthy controls will be recruited as well as 17 PTSD patients for each of the two treatment group.In terms of perspectives, this study would help isolate neural systems functionally involved in PTSD and its treatment. A better knowledge of those mechanisms would set room for the optimization of the current PTSD treatment.

ELIGIBILITY:
Inclusion Criteria:

* French speakers
* Not hospitalized grown-up patients suffering from a post-traumatic stress disorder ( PTSD) connected to one event.
* Subjects Controls: grown-up, mated with the patients in age (18 - 50 years; 4 years maximum of difference of age between a patient and his control), in sex and educational level (schooling of the 3rd level, at the level Bac+8; 3 years maximum of difference of educational level between a patient and his control)

Exclusion Criteria:

* Pregnancy
* Feeding
* Nobody under guardianship and grown-up persons being the object of a legal protective measure or not able to express their assent
* Alcoholic or addicted to drugs (including medicines)
* Other neurological disorders or psychiatric that post-traumatic stress disorder (for patients)
* Claustrophobia and contraindications in the IRMf
* Subjects controls, no known psychiatric or neurological pathology, as well as no psychiatric history.
* Persons private of freedom by a court or administrative order, persons hospitalized without assent
* Unability to read French

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2009-04; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To verify the hypothesis of a levying of inhibition of the CPFm on the tonsil, in the PTSD | 3 years

SECONDARY OUTCOMES:
Studies of the peripheral, cognitive and central mechanisms, before, then 1 week and 6 months after treatment by CBT or EMDR | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique-Hopitaux de Marseille, Marseille, France